CLINICAL TRIAL: NCT03423758
Title: Investigating the Genetic Basis of Pseudoexfoliation Syndrome, Angle-closure Glaucoma and Primary Open-angle Glaucoma
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Other Study IDs: OPHT-271016
Record Dates: First submitted 2018-01-08; First posted 2018-02-06 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma
Keywords: Pseudoexfoliation Glaucoma, Angle block glaucoma, Primary Open-Angle Glaucoma, Genetic
MeSH Terms: conditions — Glaucoma; Exfoliation Syndrome; Glaucoma, Open-Angle | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy controls: Healthy subjects with age more than 60 years
  Interventions: Other: Blood sample
- Pseudoexfoliation Glaucoma: Already diagnosed Pseudoexfoliation glaucoma patients with age more than 50 years
  Interventions: Other: Blood sample
- Angle closure Glaucoma: Already diagnosed Angle closure Glaucoma patients with age more than 21 years
  Interventions: Other: Blood sample
- Primary open-angle Glaucoma: Already diagnosed primary open-angle glaucoma with age more than 30 years
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample

SUMMARY:
There is increasing evidence that there are genetic risk factors for several forms of glaucoma, such as glaucoma caused by pseudoexfoliation syndrome (PXF) ,primary angle closure glaucoma (PACG) and primary open-angle glaucoma (POAG). The aim of the present prospective, multi-center, case-control study is to identify susceptibility genes/loci for PXF, PACG and POAG using a whole genome association (WGA) approach.

DETAILED DESCRIPTION:
As worldwide populations become older because of shifts in demography, PXF may become a matter of greater concern. The search for genes responsible for PXF may lead to the identification of key molecules in pathways critical to the normal functioning of the eye. A better understanding of normal eye function may in turn lead to more accurate diagnosis and prognosis of ocular development, and inevitably to the emergence of novel classifications based on knowledge of the molecular pathology. Such knowledge may lead to more rational disease classification, better diagnostic tests, and improved prognostic accuracy. This is of particular relevance to PXF since there is a shortage of early reliable diagnostic tests and much evidence that the early commencement of treatment can arrest progressive asymptomatic loss of vision due to PXF-related glaucoma.

The search for genes responsible for PACG may lead to the identification of key molecules in pathways critical to the normal development of the eye. A better understanding of eye development may in turn lead to more accurate diagnosis and prognosis of ocular development, and inevitably to the emergence of novel classifications based on knowledge of the molecular pathology. Such knowledge may lead to more rational disease classification, better diagnostic tests, and improved prognostic accuracy. This is of particular relevance to glaucoma since there is a shortage of early reliable diagnostic tests and much evidence that the early commencement of treatment can arrest progressive asymptomatic loss of vision for which the disease is renowned.

Identification of responsible genes for POAG development can on one hand broaden our knowledge on disease pathophysiology and on the other hand open new doors in the search for pharmacological disease modification. Especially the latter is urgently needed as IOP has for many years been the only pharmacological target and fails to prevent disease progression in a certain proportion of POAG patients.

ELIGIBILITY:
Inclusion Criteria:

1. For patients with PXF:

   * Patients with confirmed pseudoexfoliation syndrome (exfoliation glaucoma / pseudoexfoliation of the lens) in the medical history
   * Informed consent
   * Age 50 years or more
2. For patients with PACG:

   * Patients with confirmed acute primary angle closure (PAC) or primary angle closure glaucoma (PACG) in the medical history
   * Informed consent
   * Age 21 years or more
3. For healthy controls:

   * No evidence of PXF, glaucoma or uveitis during clinical examination or in the medical history
   * No evidence of major ocular disease such as diabetic retinopathy, age related macular degeneration or conditions with genetic background during clinical examination or in the medical history
   * Age more than 60 years
   * Informed consent
4. For patients with POAG:

   * Patients with confirmed primary open angle glaucoma (POAG)
   * No evidence of exfoliation glaucoma / pseudoexfoliation of the lens or pigment glaucoma
   * Informed consent
   * Age 30 or more

Exclusion Criteria:

* Patients and subjects will be excluded if one or more of the following criteria apply:
* Neovascular glaucoma
* Active or history of uveitis
* Secondary angle closure such as neovascular glaucoma or uveitis/inflammatory eye disease
* Inability to give informed consent

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal Healthy group
  2. Patients with Pseudoexfoliation Glaucoma
  3. Patients with Angle closure Glaucoma
  4. Patients with Primary open-angle Glaucoma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Genetic markers | 1 day
  To identify the genetic markers in a whole genome association screen which show very strong association with PXF, ACG and POAG. The genomic regions identified from the above analyses will be analyzed using high density single nucleotide polymorphism (SNP) chips and/or sequencing of positional candidate genes to identify causal variants.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided